CLINICAL TRIAL: NCT01407757
Title: Pharmacogenetics of Gemtuzumab Ozogamicin (GO) Therapy in Acute Myeloid Leukemia
Brief Title: Study of Gemtuzumab Ozogamicin Therapy in DNA Samples From Patients With Acute Myeloid Leukemia Treated on COG-AAML0531
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B10; COG-AAML11B10 (Other: Children's Oncology Group); AAML11B10 (Other: Children's Oncology Group); NCI-2011-03802 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-30; First posted 2011-08-02 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies; adult acute basophilic leukemia; childhood acute basophilic leukemia; adult acute eosinophilic leukemia; childhood acute eosinophilic leukemia; adult acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia without maturation (M1); adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); childhood acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute erythroleukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Gene Expression Profiling; Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene expression analysis
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: DNA analysis of blood and tissue samples may help doctors predict how well patients will respond to treatment. It may also help doctors learn more about how gemtuzumab ozogamicin works in the body.

PURPOSE: This research study is looking at gemtuzumab ozogamicin in DNA samples from patients with acute myeloid leukemia treated on COG-AAML0531.

DETAILED DESCRIPTION:
OBJECTIVES:

* To genotype the genomic DNA from acute myeloid leukemia (AML) patients treated on COG-AAML0531 clinical trial for CD33 (and PgP and SOC3) single nucleotide polymorphisms (SNPs).

OUTLINE: Archived DNA samples are analyzed for single nucleotide polymorphisms in CD33, PgP, and SOC3 genes by Sequenome platform. Results are then compared with patients clinical outcomes, including minimal-residual disease levels post induction I (chemotherapy and gemtuzumab ozogamicin), complete remission rates, refractory disease with various levels of bone marrow blasts, development of CNS/persistent disease, event-free survival, overall survival, and toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with acute myeloid leukemia
* DNA samples from patients treated on COG-AAML0531

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosed with acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Genetic changes in CD33 impact outcome of gemtuzumab ozogamicin-based therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jatinder Lamba, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota

REFERENCES:
- [Derived] Pollard JA, Guest E, Alonzo TA, Gerbing RB, Loken MR, Brodersen LE, Kolb EA, Aplenc R, Meshinchi S, Raimondi SC, Hirsch B, Gamis AS. Gemtuzumab Ozogamicin Improves Event-Free Survival and Reduces Relapse in Pediatric KMT2A-Rearranged AML: Results From the Phase III Children's Oncology Group Trial AAML0531. J Clin Oncol. 2021 Oct 1;39(28):3149-3160. doi: 10.1200/JCO.20.03048. Epub 2021 May 28. PMID 34048275
- [Derived] Tarlock K, Alonzo TA, Wang YC, Gerbing RB, Ries R, Loken MR, Pardo L, Hylkema T, Joaquin J, Sarukkai L, Raimondi SC, Hirsch B, Sung L, Aplenc R, Bernstein I, Gamis AS, Meshinchi S, Pollard JA. Functional Properties of KIT Mutations Are Associated with Differential Clinical Outcomes and Response to Targeted Therapeutics in CBF Acute Myeloid Leukemia. Clin Cancer Res. 2019 Aug 15;25(16):5038-5048. doi: 10.1158/1078-0432.CCR-18-1897. Epub 2019 Jun 10. PMID 31182436
- [Derived] Vujkovic M, Attiyeh EF, Ries RE, Goodman EK, Ding Y, Kavcic M, Alonzo TA, Wang YC, Gerbing RB, Sung L, Hirsch B, Raimondi S, Gamis AS, Meshinchi S, Aplenc R. Genomic architecture and treatment outcome in pediatric acute myeloid leukemia: a Children's Oncology Group report. Blood. 2017 Jun 8;129(23):3051-3058. doi: 10.1182/blood-2017-03-772384. Epub 2017 Apr 14. PMID 28411282